CLINICAL TRIAL: NCT05670327
Title: Diaphragmatic Dysfunction Predicts Difficult Weaning From Mechanical Ventilation After Bilateral Lung Transplantation: a Prospective Clinical Study.
Brief Title: Diaphragmatic Ultrasound and Weaning After Lung Transplant.
Status: Completed | Type: Observational
Sponsor: University of Padova (Other)
Responsible Party: Principal Investigator, Annalisa Boscolo, Principal investigator, University of Padova
Other Study IDs: LUS_BLT
Record Dates: First submitted 2022-08-28; First posted 2023-01-04 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2022-12

CONDITIONS: Diaphragm; Diaphragm Disease; Diaphragm Issues; Weakness, Muscle
Keywords: bilateral lung transplant; diaphragmatic dysfunction
MeSH Terms: conditions — Muscle Weakness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Bilateral lung recipients: Adult patients undergoing bilateral LT, not requiring invasive mechanical ventilation before surgery, were eligible for inclusion in the study only when they met the predefined 'readiness-to-wean' criteria on daily screening and were therefore deemed ready to undergone a first 30-min weaning trial.
  Interventions: Other: Diaphragmatic ultrasound assessment

INTERVENTIONS:
Other: Diaphragmatic ultrasound assessment — TFdi, diaphragmatic dysplacement, NAVA assessment, respiratory paramenters

SUMMARY:
The prevalence and adverse effect of diaphragm dysfunction (DD) after bilateral-lung transplant (LT) are still unclear, despite a well-known negative impact on weaning and outcome in other cohorts of critically ill and surgical patients.

Objects: The primary aim is investigating the prevalence of DD, assessed using point-of-care ultrasound and defined as diaphragm thickening fraction (TFdi) < 29%, at the first weaning trial after LT.

Secondary aims are investigating the impact of DD on weaning (defined success or failure according to pre-defined criteria, neuroventilatory efficiency (EAdi or NVE), perioperative (14-day) pneumonia, ICU length of stay (LOS), in-hospital mortality, and identifying potential risk factors for DD. Moreover, we aim to study the correlation between TFdi versus EAdi/NVE and the rapid shallow breathing index (RSBI), respectively.

DETAILED DESCRIPTION:
This is a prospective observational cohort study, approved by the Institutional Ethical Committee of Padua (reference number AOP2722). Written informed consent was obtained from each patient during the preoperative visit. All consecutive LT patients admitted to the Intensive Care Unit of the University Hospital of Padua were screened. Adult patients undergoing bilateral LT, not requiring invasive mechanical ventilation before surgery, were eligible for inclusion in the study only when they met the predefined 'readiness-to-wean' criteria on daily screening and were therefore deemed ready to undergone a first 30-min weaning trial. Exclusion criteria were: presence of neuromuscular blockers in the previous 12 hours, lack of ultrasound acoustic window, decline to participate, right hemi-diaphragmatic palsy due to surgical sacrifice of right phrenic nerve, duplicated patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients
* bilateral LT
* absent invasive mechanical ventilation before surgery
* fullfilling 'readiness-to-wean' criteria on daily screening (and therefore deemed ready to undergone a first 30-min weaning trial)

Exclusion Criteria:

* presence of neuromuscular blockers in the previous 12 hours
* lack of ultrasound acoustic window
* decline to participate
* right hemi-diaphragmatic palsy due to surgical sacrifice of right phrenic nerve
* duplicated patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Bilateral lung transplant at the first graft.
Sampling Method: Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2021-06-22 (Actual); Primary Completion 2022-10-19 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Diaphragmatic dysfunction at ultrasound assessment | through study completion, an average of 1 yea
  Prevalence of DD, assessed using point-of-care ultrasound and defined as diaphragm thickening fraction (TFdi) < 29% at the first weaning trial after lung transplant

SECONDARY OUTCOMES:
Impact of TFdi on weaning | through study completion, an average of 1 year
  the impact of DD, assessed using TFdi, on weaning (defined simple, difficult or prolonged according to pre-defined criteria).
Relevant clinical correlation (spearman correlation) | through study completion, an average of 1 yea
  Searman correlation between TFdi and neuroventilatory efficiency (NVE) and between TFdi and rapid shallow breathing index (RSBI)
Relation between invasive mechanical ventilation (IMV) before the first weaning trial and TFdi | through study completion, an average of 1 yea
  nonlinear correlation between IMV and TFdi

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Anaesthesia and Intensive Care, Padua University hospital, Padua, Italy

IPD SHARING:
Plan to Share IPD: No